CLINICAL TRIAL: NCT04936399
Title: Clinical Characteristics, Outcomes and Quality of Life in Patients With Squamous Cell Oesophageal Carcinoma Receiving Nivolumab After Prior Chemotherapy as Part of an Early Access to Medicines Scheme (EAMS) Program in the United Kingdom
Brief Title: A Study of Participants With Squamous Cell Oesophageal Carcinoma Receiving Nivolumab as Part of an Early Access to Medicines Scheme (EAMS) Program in the United Kingdom
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-76A
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: BMS-936558; Early Access to Medicines Scheme; EAMS; Nivolumab; Prospective Study; Quality of Life; Real World Evidence; Squamous Cell Oesophageal Carcinoma; Survival
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with Squamous Cell Oesophageal Carcinoma Receiving Nivolumab
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Participants will receive Nivolumab after prior chemotherapy as part of an early access to medicines scheme (EAMS) program in the United Kingdom (UK)
  Other Names: Opdivo®, BMS-936558

SUMMARY:
This purpose of this observational study is to review medical chart and patient survey data collection within an early access to medicines scheme (EAMS) program. Participant who are eligible, provide consent and enroll into the squamous cell oesophageal cancer EAMS to receive Nivolumab will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (≥18 years of age) enrolling into the squamous cell (including adenosquamous) oesophageal cancer early access to medicines scheme (EAMS) and plans to initiate treatment with nivolumab
* Willing and able to comply with the study requirements and provide informed consent

Exclusion Criteria:

• Does not receive at least one dose of nivolumab as part of the EAMS

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study consisting of medical chart review and patient survey data collection within an early access to medicines scheme (EAMS) program. Participants who are eligible, provide consent and enroll into the squamous cell oesophageal Cancer EAMS to receive nivolumab will be included in this study. The total number of patients and sites will be dependent on the number of requests for patient enrolment submitted to BMS from physicians. Pseudo-anonymized data on patient and disease characteristics, medical and oesophageal cancer treatment history, and nivolumab treatment patterns will be collected from patient medical charts and entered into an electronic data capture (EDC) system.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Age | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Gender | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Race | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Eastern Cooperative Oncology Group Performance Status (ECOG PS) | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Condition which the product is being used for | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Number of organs with metastases | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Sites of metastasis | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Prior surgery for oesophageal cancer | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Underlying comorbidities | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Concomitant medication | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Weight | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Disease history | At baseline
Distribution of demographic characteristics of NSCLC participants treated with nivolumab at initiation of nivolumab treatment: Treatment history | At baseline
Distribution of treatment patterns of nivolumab: Treatment duration | Up to 12 months
Distribution of disease progression to determine progression free survival (PFS) based on data collected as part of routine care | Up to 12 months
Distribution of disease progression to determine overall survival (OS) based on data collected as part of routine care | Up to 12 months
Distribution of survival status to determine progression free survival (PFS) based on data collected as part of routine care | Up to 12 months
Distribution of survival status to determine overall survival (OS) based on data collected as part of routine care | Up to 12 months
Distribution of patient quality of life through EQ-5D-3L (EQ-5D) at baseline following patient enrolment into the EAMS | At baseline
Distribution of patient quality of life through EQ-5D-3L (EQ-5D) every two weeks for 24 weeks post-treatment initiation following patient enrolment into the EAMS | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United Kingdom (33):
  - Local Institution - 0006, Truro, Cornwall
  - Local Institution, London, Greater London
  - Local Institution, Maidstone, Kent
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Grimsby, Lincolnshire
  - Local Institution, Edinburgh, Scotland
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Leeds, West Yorkshire
  - Local Institution, Basingstoke
  - Local Institution, Bebington
  - Local Institution, Belfast
  - Local Institution, Birmingham
  - Local Institution, Blackburn
  - Local Institution - 0037, Bristol
  - Local Institution, Cambridge
  - Local Institution, Cardiff
  - Local Institution, Cottingham
  - Local Institution, Coventry
  - Local Institution, Derby
  - Local Institution, Devon
  - Local Institution, Dundee
  - Local Institution, Headington
  - Local Institution, Lancaster
  - Local Institution, London
  - Local Institution, Manchester
  - Local Institution, Melrose
  - Local Institution, Northwood
  - Local Institution, Nottingham
  - Local Institution, Pembrokeshire
  - Local Institution, Preston
  - Local Institution, Surrey
  - Local Institution, Taunton
  - Local Institution, Walsall

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Pre-approval Access (PAA) Healthcare Practitioner Requests — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine/investigational-drugs-available.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome